CLINICAL TRIAL: NCT05334056
Title: Drug Test Detection 24 Hours After Nasal Administration of Cocaine as a Local Vasoconstrictor Prior to Nasal Intubation
Brief Title: Drug Test Detection of Cocaine for Nasal Intubation
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mo Haslund Larsen, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: 50510617; 2021-000709-26 (EudraCT Number); H-21028055 (Other: Regional Committee on Health Research Ethics)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cocaine Adverse Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and whole blood samples.
  Saliva samples will be analyzed immediately following collection and disposed as biological waste upon securing the analysis result.
  Whole blood samples will be stored until inclusion is complete and will hereafter be analyzed in one batch. Immediately following analysis the samples will be discarded as biological waste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cocaine Nasal — 2 ml of 4% cocaine given as a nasal spray immediately prior to nasal intubation
  Other Names: Cocaine 4%

SUMMARY:
The objective of this study is to determine whether it is possible to detect traces above national cut-offs of either cocaine's main metabolite benzoylecgonine in saliva or cocaine in blood 24 hours after administering 2 ml of 40 mg/ml cocaine-saline to the nasal mucosa.

The investigators hypothesize that the level of cocaine's main metabolite bezoylecgonine in saliva after cocaine administered for anesthetic purposes will be below detection limits after 24 hours.

DETAILED DESCRIPTION:
When performed by trained personnel nasotracheal intubation is a safe and effective technique for attaining a secure airway in preparation for surgery of the head and neck. Prior to nasal intubation the mucosa must be sufficiently lubricated and decongested in order to minimize epistaxis. When intubation is performed on awake patients anesthesia of the nose is also necessary. Cocaine has for many years been used for both decongestive and anesthetic purposes due to its unique pharmacodynamic profile. When applied to the nasal mucosa its vasoconstrictive quality aids in facilitating the inspection of the nasal cavity whilst the anesthetic effect allows for manipulation within the cavity. The vasoconstriction arises through cocaine's ability to inhibit the reuptake and metabolism of catecholamines, which then in greater concentration has adrenergic effects. By binding to and blocking axonal membrane sodium channels, cocaine interferes with the propagation of action potentials and thereby also exerts an analgesic effect.

Along with other countries Denmark has a legal zero tolerance policy for a long list of drugs in drivers including cocaine. During routine screenings or if the police suspect a driver to be under the influence of illegal drugs, they will first complete a qualitative saliva analysis testing for cocaine's main metabolite benzoyelecgonine. If the test comes out positive or there are clinical signs of drug influence, a supplementary blood sample measuring cocaine will be drawn and analyzed for use in the legal system. Repercussions from a cocaine test value exceeding the legal limit consists of a large fine, driver's license revocation and mandatory participation in a drug and alcohol course, neither of which seems fair to inflict on the uninformed and consequently unaware patient.

Pharmacokinetics for nasal cocaine have been described but no studies defining proper instructional driving precautions appear to exist. One study recommended patients be informed and consent prior to cocaine administration and be warned they may fail a drug test up to 72 hours postoperatively but as of 2021 patients are in many countries - including Denmark - still not informed about this time limit.

When administered in doses thought to avoid systemic effects, cocaine is a safe local anesthetic agent. The recommended dosage varies considerably throughout the literature with safe doses ranging between 1.5-3.0 mg/kg. The amount of cocaine absorbed has in one study been found to be 5% but has not been subsequently verified. The dosage of cocaine used prior to nasal intubation in Denmark is typically 1-2 ml of 4% cocaine resulting in a total dose of 40-80 mg. The typical 'street dose' is 40-100 mg. The Danish cut-off values for detection of cocaine's main metabolite benzoylecgonine is 200 ng/ml in saliva and 0.01 mg/kg in whole blood.

The investigators wish to evaluate whether cocaine levels exceed detection limits 24 hours after administration prior to nasal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for nasal intubation
* Proficient in spoken and written Danish
* Negative baseline cocaine saliva test

Exclusion Criteria:

* Intubation to be done on awake patient
* Pregnancy

  * Women of childbearing potential must produce a negative hCG urine stix to participate
* Known symptomatic coronary artery disease

  * As declared by patient or noted in the patient's file
* Untreated hypertension

  * As declared by patient or noted in the patient's file
  * Not taking antihypertension drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients schedualed to undergo surgery at Rigshospitalet with the use of nasal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Saliva analysis | 24 hours after cocaine administration
  Analysis of cocaine's main metabolite benzoylecgonine in saliva measured in nanograms per milliliter

SECONDARY OUTCOMES:
Whole blood toxicology | 1 hour and 24 hours after cocaine administration
  Analysis of cocaine in a whole blood sample measured in nanograms per milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Mo Haslund Larsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No